CLINICAL TRIAL: NCT03861546
Title: Better Together: Leveraging Primary Care and Social Network Resources to Create a Patient-centered Approach to Improve Diabetes Among South Asians
Brief Title: Developing a Lifestyle Intervention for South Asians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Megha Kumudchandra Shah, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00097724
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Behavior, Health; Pre Diabetes; Diabetes
Keywords: South Asian adults; Patient-centered approach; Intensive lifestyle interventions; Diabetes
MeSH Terms: conditions — Health Behavior; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy lifestyle Shared Medical Appointment (SMA) program (Experimental): South Asian (SA) adults with prediabetes and Type 2 Diabetes (T2D) that are 'information rich' and have variation in background characteristics will be identified. Dyads (spouses, parent/adolescent or young adult child, peers) will participate in a 16-week culturally-tailored, community-informed pre-post SMA intervention to improve health behaviors.
  Interventions: Behavioral: Healthy lifestyle Shared Medical Appointment (SMA) program

INTERVENTIONS:
Behavioral: Healthy lifestyle Shared Medical Appointment (SMA) program — Social network-based, culturally-tailored healthy lifestyle SMA program for high risk SAs will be piloted to collect pre-post data on diet and exercise habits, and to determine feasibility and acceptability. Patients will participate in physician-led group visits every other week focused on improving dietary and exercise practices to reduce weight. Biometric measurements (weight, height, blood pressure) will be collected, point of care glucose and lipid testing will be done.

SUMMARY:
This study aims to test the hypothesis that a culturally tailored lifestyle intervention can improve health behaviors among South Asians with prediabetes and diabetes

DETAILED DESCRIPTION:
This pre-post pilot study is a 16 week lifestyle program for South Asians with prediabetes or diabetes in Atlanta. Patients will participate in physician-led group visits every other week focused on improving dietary and exercise practices to reduce weight.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years;
2. confirmed diagnosis of prediabetes or T2D (documented A1c of ≥ 5.7%, 2-hour post-load glucose of >140, or FBG of >100);
3. a family member or peer willing to participate and attend all sessions as a social influencer;
4. proficiency in English of at least one member of each dyad,
5. willingness to provide written consent.

Exclusion Criteria:

1. type 1 diabetes or diabetes secondary to other conditions (e.g. steroid-induced, pancreatic insufficiency, or chemotherapy-induced);
2. malignancy or life-threatening illness with life expectancy of <5 years;
3. end-stage disease or serious illness that prohibits participation (e.g. end-stage renal disease or class IV congestive heart failure);
4. inability to perform unsupervised physical activity;
5. pregnancy;
6. diagnosed cognitive deficits or limited decision-making capacity;
7. alcohol or substance abuse;
8. homelessness or no fixed address.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-03-03 (Actual); Primary Completion 2019-06-23 (Actual); Study Completion 2019-06-23 (Actual)

PRIMARY OUTCOMES:
Participant perceptions of SMA program | 4 months
  Physician-participants interviews will be digitally audio-recorded and transcribed verbatim, with de-identified transcripts analyzed.
SMA program retention rate | 4 months
  Number of participants retained will be recorded and SMA retention rate will be calculated

SECONDARY OUTCOMES:
Change in body mass index (BMI) | Baseline, 4 months, and 12 months
  Body Mass Index (BMI) is a number representing person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
Change in blood pressure | Baseline, 4 months, and 12 months
  Blood pressure will be measured pre- and post- intervention
Change in blood cholesterol level | Baseline, 4 months, and 12 months
  Cholesterol level will be measured by blood test pre- and post- intervention
Change in physical activity daily minutes | Baseline, 4 months, and 12 months
  Daily minutes of moderate intensity exercise will be self reported by participants
Change in step counts | Baseline, 4 months, and 12 months
  Daily step counts (using wearable perdometer) will be recorded.
Change in diet | Baseline, 4 months, and 12 months
  Pre-post assessment of change in consumption will be done using food frequency questionnaire. It has 16 questions that assess dietary habits over the past week.

CONTACTS AND LOCATIONS:
Overall Officials: Megha K Shah, MD, Principal Investigator — Emory University
Locations (1):
- Emory Family Medicine Clinic, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah MK, Naing S, Kurra N, Weber MB, Islam N, Ali MK, Narayan KMV. A culturally adapted, social support-based, diabetes group visit model for Bangladeshi adults in the USA: a feasibility study. Pilot Feasibility Stud. 2022 Jan 24;8(1):18. doi: 10.1186/s40814-022-00974-9. PMID 35074000